CLINICAL TRIAL: NCT06283836
Title: Dexmedetomidine Continuous Intravenous Infusion vs. Remifentanil Target-controlled Infusion Conscious Sedation for Stapedotomy/Stapedectomy- a Prospective, Single-center, Double-masked Randomized Trial
Brief Title: Dexmedetomidine vs. Remifentanil Conscious Sedation for Stapedotomy/Stapedectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Breazu Caius Mihai, MD, PhD, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Dexrem ATI 4-6
Record Dates: First submitted 2024-02-14; First posted 2024-02-28 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-08

CONDITIONS: Otosclerosis
Keywords: otosclerosis; dexmedetomidine; remifentanil; sedation; satisfaction score
MeSH Terms: conditions — Otosclerosis | interventions — Dexmedetomidine; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients and surgeons were blinded to the group allocation and the personnel providing postoperative care and collecting the postoperative data were also unaware of the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group D (Active Comparator): Continuous infusion of dexmedetomidine during intervention ( 1ug/kg over 15 minutes then 0.4 ug/kg/hour)
  Interventions: Drug: Dexmedetomidine
- Group R (Active Comparator): Target-controlled infusion of remifentanil ( 2ng//ml- plasma concentration)
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Dexmedetomidine — monitored anesthesia care (sedation)
  Arms: Group D
Drug: Remifentanil — monitored anesthesia care (sedation)
  Arms: Group R

SUMMARY:
Dexmedetomidine continuous intravenous infusion vs. remifentanil target-controlled infusion conscious sedation for stapedotomy/stapedectomy- a prospective, single-center, double-masked randomized trial

The goal of this clinical trial is to compare monitored anesthesia care with continuous intravenous dexmedetomidine vs. remifentanil target-controlled infusion in patients undergoing stapedotomy or stapedectomy for otosclerosis. The aims of this research are:

* to assess the patient's satisfaction with each sedation regimen
* the surgeon will also grade their satisfaction regarding the surgical field The investigators will monitor and analyze the vitals during and after the intervention and document any intra- and postoperative complications.

Participants will be randomly assigned to receive either dexmedetomidine or remifentanil, and the patient, the surgeon, and other care providers except the attending anesthesiologist will not be aware of the treatment administered.

DETAILED DESCRIPTION:
Otosclerosis has a disabling character through progressive hearing reduction. The etiopathogenetic process consists of osteodystrophy degeneration of the otic capsule, leading to decreased mobility of the stapes bone of the middle ear and causing conductive or mixed hearing loss. It is relatively common in ENT (ear, nose and throat) pathology, generally affecting young adults with a 4:1 ratio between women and men. Treatment is surgical by stapedotomy or stapedectomy and placement of a Teflon prosthesis designed to restore the vibratory capacity of the ossicular complex of the middle ear. Anesthetic management consists, depending on institutional custom, surgeon, or patient preference, in general anesthesia or, relatively frequently, monitored anesthesia care alongside local anesthesia. There is no specific regional anesthesia technique for middle ear interventions because the ear exhibits heterogeneous sensory innervation containing branches from the cervical plexus and cranial nerves V, VII, and X. Local anesthesia consists of circular infiltration of the ear canal and association with an effective sedation technique is indispensable for patient and operator comfort. The objectives of sedation are:

* An immobile operating field.
* Minimal bleeding.
* Hemodynamic and respiratory stability.
* Reducing the risk of postoperative nausea and vomiting.
* Patient comfort. The significant advantage of conscious sedation over general anesthesia or deep sedation is the possibility of real-time feedback from the patient in case of vertigo or for hearing testing after fitting the prosthesis. Deep sedation may also produce an uncooperative patient with involuntary movements or upper airway obstruction under conditions of problematic access to the cephalic extremity that may compromise the operating field.

Dexmedetomidine is a selective alpha-2 adrenergic receptor agonist that appeared in clinical anesthetic practice relatively recently, with sedative effects, reduction of required opioid doses, reduced frequency of delirium and agitation, perioperative sympathicolysis, cardiovascular stabilizing impact and preservation of respiratory function.

Remifentanil is a synthetic, potent, ultrashort-lived opioid used for postoperative analgesia, sedation, or general anesthesia.

The objective of this study is to compare dexmedetomidine (continuous infusion) to remifentanil (target-controlled infusion according to the Minto model) for monitored anesthesia care of a cohort of patients with otosclerosis presenting for stapedectomy/stapedotomy at the ENT Clinic - Cluj County Clinical Emergency Hospital.

ELIGIBILITY:
Inclusion Criteria:

* otosclerosis surgery, ASA ( American Society of Anesthesiologists) status 1-2

Exclusion Criteria:

* ASA status 3-4
* requiring general anesthesia
* refusing to participate
* allergic to study medication
* severe bradicardia, atrioventricular block
* cognitive impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 24 hours
  Iowa Satisfaction with Anaesthesia Scale after full recovery. Range between -3 (poor satisfaction) to +3 (very satisfied)
Surgeon satisfaction | Immediately after procedure
  Surgeon satisfaction score to be assessed on a 1-4 VAS after the procedure ( 1-poor, 2-moderate, 3-good, 4-excellent)

SECONDARY OUTCOMES:
mean arterial pressure | 6 hours
  the variation of blood pressure during intervention and postoperative
Heart Rate | 6 hours
  Heart rate variation during intervention and postoperative

OTHER OUTCOMES:
the need for adjuncts during intervention | during surgery
  insufficient sedation grade or analgesia requiring administration of hypnotics or opioids beyond the protocol to maintain an adequate level of comfort for patient and surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Caius Mihai Breazu, MD, PhD, Principal Investigator — Iuliu Hatieganu University of Medicine snd Pharmacy
Locations (1):
- Cluj County Clinical Emergency Hospital, Cluj-Napoca, Cluj, Romania